CLINICAL TRIAL: NCT01069328
Title: Study of BAY43-9006 (Sorafenib) in Combination With Carboplatin, Paclitaxel and Bevacizumab in Previously Untreated Patients With Stage IIIB (With Malignant Pleural Effusions) or Stage IV Non-small Cell Lung Cancer (NSCLC)
Brief Title: Dose Escalating Study With BAY43-9006 With Carboplatin, Paclitaxel and Bevacizumab in Untreated Stage IIIb Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11956
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Cancer
Keywords: Lung; cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — Sorafenib; Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006); Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin
- Arm 2 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006); Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin
- Arm 3 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006); Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin
- Arm 4 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006); Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin
- Arm 5 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006); Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin
- Arm 6 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006); Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) — Sorafenib 200 mg orally BID interrupted dosing
  Arms: Arm 1; Arm 2
Drug: Nexavar (Sorafenib, BAY43-9006) — Sorafenib 400 mg orally BID interrupted dosing
  Arms: Arm 3; Arm 4; Arm 5; Arm 6
Drug: Bevacizumab — Bevacizumab 2.5 mg/kg intravenously
  Arms: Arm 3
Drug: Bevacizumab — Bevacizumab 5 mg/kg intravenously
  Arms: Arm 1; Arm 4
Drug: Bevacizumab — Bevacizumab 7.5 mg/kg intravenously
  Arms: Arm 5
Drug: Bevacizumab — Bevacizumab 10 mg/kg intravenously
  Arms: Arm 2; Arm 6
Drug: Paclitaxel — Paclitaxel 200 mg/m² intravenously
Drug: Carboplatin — Carboplatin AUC 6 intravenously

SUMMARY:
To determine the tolerability, maximum tolerated dose and pharmacokinetics of this drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Stage IIIB (with malignant pleural effusions) or Stage IV histological or cytological confirmation of non-small cell carcinoma (excluding squamous)
* Age >/= 18 years old
* Patients must have at least 1 evaluable lesion. Lesions must be evaluated by CT scan or MRI
* ECOG Performance Status of 0 to 1
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of first dose:

  * Hemoglobin >/= 9.0 g/dL
  * White blood cell (WBC) count >/= 2,500/mm3
  * Absolute neutrophil count (ANC) >/= 1,500/mm3
  * Platelet count >/= 100,000/mm3
  * Total bilirubin </= 1.5 times the upper limit of normal (ULN)
  * ALT and AST </= 2.5 X ULN (</= 5 X ULN for patients with liver involvement)
  * INR </= 1.5 and aPTT within normal limits
  * Serum creatinine </= ULN or creatinine clearance (CrCl) >/= 45 mL/min (CrCl = Wt (kg) x (140-age)/72 x Cr level, female x 0.85) for patients with creatinine levels above institutional normal
  * Urinalysis (UA) must show less than 1+ protein in urine, or the patient will require a repeat UA. If repeat UA shows 1+ protein or more, a 24 hour urine collection will be required and must show total protein </= 1000 mg/24 hour to be eligible

Exclusion Criteria:

* Patients with squamous histology
* Cardiac disease: Congestive heart failure > Class II NYHA; active coronary artery disease (MI more than 6 months prior to study entry is allowed); or serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management
* HIV infection or chronic hepatitis B or C
* Active clinically serious infections (> Grade 2 NCI-CTC Version 3.0)
* Evidence or history of CNS disease, including primary brain tumors, seizures disorders, or any brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-07; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to define the safety profile and maximum tolerated dose (MTD) of BAY43-9006 (sorafenib) administered in combination with, carboplatin, paclitaxel and bevacizumab | 2 years

SECONDARY OUTCOMES:
The secondary objectives include evaluation of pharmacokinetics, biomarkers, pharmacodynamics and tumor response of patients treated with BAY43-9006 (sorafenib) in combination with bevacizumab, paclitaxel and carboplatin | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Rochester, Minnesota
  - Houston, Texas